CLINICAL TRIAL: NCT07090824
Title: Subcutaneous Pharmacokinetic Evaluation of Monomeric Insulin and Lyumjev in Adults With Type 1 Diabetes
Acronym: SPEED
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Rayhan A. Lal, Assistant Professor of Medicine & Pediatrics, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 71030; 2R56DK119254-06 (NIH)
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 1; Type 1 Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 1; T1D; Insulin-Dependent Diabetes Mellitus; Pharmacokinetics; Insulin; Subcutaneous Insulin; Drug: Insulin Lispro; Drug: Insulin Regular; Drug: Modified Insulin Formulations; Drug: Insulin Lispro-aabc; Insulin formulation; Monomeric Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Randomized, three-period, three-treatment crossover study. Each participant will receive all three insulin formulations (diluted U-200 Humalog, diluted U-500 Humulin, and U-100 Lyumjev) in randomized sequence across three separate visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Diluted Humalog U-200 Insulin (Experimental): Participants will receive 0.20u/kg U-200 Humalog diluted 1:1 with sterile water, EDTA, and mannitol dilution buffer (final concentration U-100) through subcutaneous injection
  Interventions: Drug: Diluted Humalog U-200 Insulin; Dietary Supplement: Boost Mixed Meal Test
- Diluted Humulin U-500 Insulin (Experimental): Participants will receive 0.20u/kg U-500 Humulin diluted 1:4 with sterile water, EDTA, and mannitol dilution buffer (final concentration U-100) through subcutaneous injection
  Interventions: Drug: Diluted U-500 Humulin Insulin; Dietary Supplement: Boost Mixed Meal Test
- Lyumjev U-100 Insulin (Active Comparator): Participants will receive 0.20 u/kg commercially available U-100 Lyumjev insulin (unmodified) through subcutaneous injection.
  Interventions: Drug: Lyumjev U-100 Insulin; Dietary Supplement: Boost Mixed Meal Test

INTERVENTIONS:
Drug: Diluted Humalog U-200 Insulin — Commercially available U-200 Humalog (insulin lispro) diluted 1:1 with a dilution buffer composed of sterile water, EDTA and mannitol to achieve U-100 concentration. Administered as single subcutaneous injection at 0.20 u/kg body weight following mixed meal consumption.
  Arms: Diluted Humalog U-200 Insulin
Drug: Diluted U-500 Humulin Insulin — Commercially available U-500 Humulin (regular insulin) diluted 1:4 with dilution buffer composed of sterile water, EDTA and mannitol to achieve U-100 concentration. Administered as single subcutaneous injection at 0.20 u/kg body weight following mixed meal consumption.
  Arms: Diluted Humulin U-500 Insulin
Drug: Lyumjev U-100 Insulin — Commercially available U-100 Lyumjev (insulin lispro-aabc) administered unmodified as comparator. Administered as single subcutaneous injection at 0.20 u/kg body weight following mixed meal consumption.
  Arms: Lyumjev U-100 Insulin
Dietary Supplement: Boost Mixed Meal Test — Standardized mixed meal (Boost drink) administered at 8.0 mL/kg body weight (17.3 g carbohydrates per 100 mL) consumed immediately before insulin injection at each visit.

SUMMARY:
The SPEED study is a randomized, crossover pilot study evaluating the pharmacokinetics of novel insulin formulations in adults with type 1 diabetes. The study compares two experimental insulin formulations (diluted U-200 Humalog and U-500 Humulin with sterile water, mannitol and EDTA) against commercially available U-100 Lyumjev to determine if these modifications can improve insulin onset and duration of action.

Twenty participants will complete three study visits, each separated by at least48 hours. At each visit, participants will receive one of the three insulin formulations (0.20 u/kg) via subcutaneous injection following consumption of a standardized mixed meal. Blood samples will be collected frequently over 6 hours to measure insulin concentrations and assess pharmacokinetic parameters, including time to maximum concentration (Tmax), maximum concentration (Cmax), elimination half-life, and area under the curve.

The study aims to address limitations of current insulin formulations used in automated insulin delivery systems, which are too slow to provide optimal meal coverage without pre-meal dosing. By reducing zinc content through EDTA chelation and decreasing metacresol concentration through dilution, these novel formulations may offer faster onset and shorter duration of action, potentially improving glucose control in people with type 1 diabetes using insulin pump therapy.

DETAILED DESCRIPTION:
Background and Rationale Current rapid-acting insulin formulations used in automated insulin delivery systems are limited by slow pharmacokinetics that prevent optimal meal coverage without pre-meal announcement. These insulins are predominantly composed of hexamers (94%) when stored, which must dissociate to monomers for biological activity. The presence of zinc ions and metacresol in commercial formulations promotes hexamer stability, contributing to slower onset and prolonged duration of action.

This study evaluates a two-pronged approach to improve insulin pharmacokinetics: (1) zinc removal through EDTA chelation, and (2) metacresol concentration reduction through dilution. Previous research has shown that these modifications can improve oligomer composition and potentially enhance insulin action speed and duration.

Study Design This is a randomized, crossover, single-dose, within-subject pilot study. Each participant serves as their own control, receiving all three insulin formulations in randomized order across three separate visits.

Target Enrollment: 10 participants

Key Inclusion Criteria

* Age 18-60 years
* Clinical diagnosis of type 1 diabetes
* Insulin pump therapy and continuous glucose monitor use for ≥3 months
* For females: not pregnant or trying to conceive
* Ability to provide informed consent and follow protocol requirements

Key Exclusion Criteria

* Diabetic ketoacidosis in past 3 months
* Severe hypoglycemia (seizure/loss of consciousness) in past 3 months
* Blood donation within 8 weeks
* Known clinically significant anemia
* Pregnancy or lactation
* Active infection
* Chronic kidney disease (GFR <60 mL/min/1.73m²)

Study Interventions

Three insulin formulations will be tested:

* Test Insulin #1: U-200 Humalog diluted 1:1 with sterile water, EDTA, and mannitol solution to achieve U-100 concentration
* Test Insulin #2: U-500 Humulin diluted 1:4 with sterile water, EDTA, and mannitol solution to achieve U-100 concentration
* Comparator: U-100 Lyumjev (commercially available, unmodified)

All formulations will be prepared by Stanford Healthcare Investigational Drug Services Pharmacy under aseptic conditions and used within 2 hours of preparation.

Study Procedures

* Pre-injection: Participants suspend insulin delivery 60 minutes before injection and consume a standardized mixed meal (Boost drink at 8.0 mL/kg body weight, providing 17.3 g carbohydrates per 100 mL).
* Injection: Subcutaneous injection of assigned insulin at 0.20 u/kg body weight.

Sample Collection:

* Frequent blood sampling (4 mL EDTA tubes) every 5 minutes for first 60 minutes, then every 15 minutes until 360 minutes.
* Real-time glucose monitoring using Contour Next One glucometer
* Early termination allowed if glucose increases after 240 minutes
* Maximum blood volume: 132 mL per visit (or 2.0 mL/kg if <66 kg)

Sample Processing:

Blood samples centrifuged immediately, plasma transferred to microcentrifuge tubes in triplicate, frozen on dry ice, and stored at -80°C until insulin ELISA analysis.

Primary Endpoints

Pharmacokinetic parameters for each insulin formulation:

* Time to maximum insulin concentration (Tmax)
* Maximum plasma insulin concentration (Cmax)
* Elimination half-life (T1/2)
* Area under the concentration-time curve (AUC)

Statistical Analysis Non-parametric methods will be used due to small sample size. The Wilcoxon signed-rank test will compare insulin formulations, with statistical significance set at p<0.05. Results will be presented as median and interquartile range for each parameter.

Safety Considerations The study is categorized as no greater than low risk.

Potential risks include:

* Standard blood draw complications (pain, bruising, bleeding)
* Hyperglycemia from mixed meal or hypoglycemia from insulin
* Transient local reactions at injection site from EDTA-containing formulations Glucose monitoring will be increased to every 5 minutes if levels fall below 70 mg/dL.

Follow-up Participants will be contacted 1-2 days after each visit to assess for unusual hypoglycemic or hyperglycemic episodes.

Future Research With participant consent, stored blood samples may be used for future approved research studies. Samples will be identified only by study ID number to maintain confidentiality.

Significance This study addresses a critical limitation in current diabetes management technology. Despite advances in automated insulin delivery systems, slow insulin pharmacokinetics leave even well-controlled patients spending 5+ hours daily outside target glucose range. If successful, these novel formulations could significantly improve glucose control and quality of life for people with type 1 diabetes using insulin pump therapy.

Study Contact Information:

Ryan Kingman, Clinical Research Coordinator Email: rkingman@stanford.edu Institution: Stanford University Office: 453 Quarry Road, Palo Alto, CA 94304

Principal Investigator:

Rayhan Lal, MD Stanford University

Study Location:

Stanford Clinical and Translational Research Unit 800 Welch Road, Palo Alto, CA

Regulatory Information:

IND Number: 169699 Funding Source: Other (Non-NIH)

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, a subject must meet all of the following criteria:

1. 18-60 years of age
2. Clinical diagnosis of type 1 diabetes
3. On insulin pump therapy and continuous glucose monitor for at least 3 months
4. For females of childbearing potential, a negative pregnancy test and not attempting to conceive.
5. Understanding and willingness to follow the protocol and sign informed consent
6. Ability to speak, read and write English

Exclusion Criteria:

The presence of any of the following is an exclusion for the study:

1. Diabetic ketoacidosis within 3 months
2. Severe hypoglycemia resulting in seizure or loss of consciousness within 3 months prior to enrollment
3. Have donated blood within 8 weeks
4. Have a known clinically significant history of anemia
5. Pregnant or lactating
6. Active infection
7. Any medical condition that, in the investigator's opinion, might interfere with study completion or participant safety.
8. Known seizure disorder
9. Inpatient psychiatric treatment within 6 months
10. Medication instability within 1 month prior to enrollment, including antihypertensive, thyroid, antidepressant, or lipid-lowering medications
11. Suspected drug or alcohol abuse
12. Chronic kidney disease (GFR < 60 mL/min/1.73m²)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Time to Maximum Insulin Concentration (Tmax) | 0 to 360 minutes post-injection
  Time from insulin injection to maximum plasma insulin concentration for each insulin formulation, determined from frequent blood sampling data. Measured using validated enzyme-linked immunosorbent assay (ELISA).
Maximum Plasma Insulin Concentration (Cmax) | 0 to 360 minutes post-injection
  Peak plasma insulin concentration achieved for each insulin formulation, determined from frequent blood sampling data. Measured using validated enzyme-linked immunosorbent assay (ELISA).
Elimination Half-Life (T1/2) | 0 to 360 minutes post-injection
  Time required for plasma insulin concentration to decrease by 50% from maximum concentration for each insulin formulation, calculated from frequent blood sampling data. Measured using validated enzyme-linked immunosorbent assay (ELISA).
Area Under the Concentration-Time Curve (AUC) | 0 to 360 minutes post-injection
  Total drug exposure calculated as the area under the plasma insulin concentration-time curve using the trapezoidal rule. Provides a weighted sum of insulin concentration values over time for each formulation. Measured using validated enzyme-linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Rayhan A Lal, MD, Principal Investigator — Stanford University; Eric Appel, PhD, Study Director — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared. Data will be made available to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  Requests should be directed to eappel@stanford.edu. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 18 months after article publication and ending 5 years following article publication.
Access Criteria: Proposals should be directed to eappel@stanford.edu. To gain access, data requestors will need to sign a data access agreement.